CLINICAL TRIAL: NCT04809077
Title: Focus on the Humeral Component Following Reverse Shoulder Arthroplasty: Radiographic and Clinical Findings
Brief Title: Focus on the Humeral Component Following Reverse Shoulder Arthroplasty
Acronym: RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S63831
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Arthropathy
Keywords: Reverse total shoulder arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reverse total shoulder replacement (Other): Patients who underwent a total shoulder replacement using a reverse type implant (Delta Xtend or Zimmer TM)
  Interventions: Other: Reverse total shoulder replacement

INTERVENTIONS:
Other: Reverse total shoulder replacement — Long-term radiographic and clinical data of patients who underwent a reverse shoulder replacement

SUMMARY:
Reverse total shoulder arthroplasty has been widely used in the treatment of rotator cuff arthropathy. Follow-up has historically focused on the glenoid component because of problems with fixation and scapular notching leading to functional failure. Since several patients have shown cortical thinning of the proximal lateral humeral cortex during follow-up, further research is recommended to evaluate the cause and clinical impact of these radiographic changes. The goal of this study is to collect long-term radiographic and clinical data in order to facilitate the identification of risk factors.

DETAILED DESCRIPTION:
Reverse total shoulder arthroplasty has been widely used in the treatment of rotator cuff arthropathy. Follow-up has historically focused on the glenoid component because of problems with fixation and scapular notching leading to functional failure. Fixation of the humeral component has evolved from cemented to mostly uncemented with diaphyseal of metaphyseal press-fit stems. Bony changes around the stem reflect the bone-implant interface; research to evaluate and interpret these changes is insufficient at this moment. Since several patients have shown cortical thinning of the proximal lateral humeral cortex during follow-up, further research is recommended to evaluate the cause and clinical impact of these radiographic changes. The goal of this study is to collect long-term radiographic and clinical data in order to facilitate the identification of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old
* Total shoulder replacement using a reverse type implant (Delta Xtend or Zimmer TM) between 2007 and 2017 in UZ Leuven
* Primary indication for surgery is rotator cuff arthropathy
* Informed consent obtained

Exclusion Criteria:

* Total shoulder replacement in post septic arthritis.
* Total shoulder replacement in post-instability arthritis.
* Revision total shoulder arthroplasty.
* Posttraumatic total shoulder arthroplasty (after failed index operation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Shoulder X-ray | up to 20 months
  To describe bony reaction at the bone-implant interface for the humeral component of a reverse shoulder arthroplasty. End-point radiographs will be compared to radiographs taken postoperatively in order to define stress shielding and/or bone resorption in the 5 humeral zones described by Nagels et al.

SECONDARY OUTCOMES:
Clinical outcome | up to 20 months
  To relate bony changes at the bone-implant interface of the humeral component of a reverse total shoulder arthroplasty to clinical outcome
Constant-Murley score | up to 20 months
  To evaluate the functional state of the shoulder in patients with shoulder complaints
Short Form 36 Health Survey Questionnaire (SF-36) | up to 20 months
  To indicate the health status and pain scales
Net Promotor Score (NPS) | one time visit
  To evaluate patient satisfaction after surgery
Anchor Question Shoulder Score | up to 20 months
  To measure the change in general daily functioning and pain symptoms after shoulder surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Debeer, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No